CLINICAL TRIAL: NCT00389142
Title: Genetic Studies in Interstitial Cystitis/Bladder Pain Syndrome (IC/BPS)
Brief Title: Identifying Genetic Causes of IC/BPS
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Catherine Brownstein, Assistant Professor of Genetics and Pediatrics, Harvard Medical School, Boston Children's Hospital
Other Study IDs: 04-11-160; 91208 (Other Grant/Funding Number: Broad Institute)
Record Dates: First submitted 2006-10-17; First posted 2006-10-18 (Estimated); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Interstitial Cystitis; Bladder Pain Syndrome
Keywords: pelvic pain; urinary frequency; painful bladder; urinary urgency
MeSH Terms: conditions — Cystitis, Interstitial; Pelvic Pain

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The investigators will collect and store DNA (via blood or saliva) and urine samples on all participants (affected and unaffected family members). Bladder tissue if available from clinical procedure will be collected in affected participants only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1 cohort: All participants will undergo genome sequencing and urinalysis studies.

SUMMARY:
Interstitial cystitis (IC), also called Bladder Pain syndrome (BPS) is a common condition with no known cause or cure. Twin studies and family accounts have suggested that the condition may be genetic or passed down (inherited) from one generation to another.

In this study, the investigators are collecting genetic material via blood or saliva and medical information from families in North America in an attempt to identify genetic factors that may cause IC/BPS. The investigators are enrolling inviduals with IC/BPS and their family members (family members with and without IC like symptoms). Travel to Boston not required.

DETAILED DESCRIPTION:
The investigators are trying to identify a genetic cause of interstitial cystitis (IC)/bladder pain syndrome (BPS). The investigators are looking to enroll individuals with a clinical diagnosis of IC/BPS and their family member. The investigators are attempting to determine if there is a connection between symptoms of IC/PBS and changes in specific genes or a pathway of connected genes. The investigators will use several genetic technologies including but not limited to; linkage analysis, genome sequencing, RNAseq and candidate gene studies to try to identify the cause of IC/BPS. Once the investigators identify the cause of IC/BPS they will be able to identify and design more effective treatments for affected individuals. The investigators are looking for families with IC/BPS symptoms to give a DNA sample (from blood/saliva), urine samples, and answer several questionnaires. Travel to Boston NOT necessary.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IC/BPS
* Males and females of any age
* Urinary frequency - more than 1X/hour, and/or
* Dysuria, and/or
* Pelvic, suprapubic, or abdominal pain - for 3 months or longer
* Nocturia
* Normal urinary stream (by history)
* No evidence of active bacterial UTI (no pyuria & negative urinary culture for last 3 months)
* First degree relative of someone with above symptoms

Exclusion Criteria:

* Major structural/anatomical urinary tract abnormalities by ultrasound
* Underlying inborn conditions affecting the urinary tract
* Surgery/chemotherapy affected pelvic area
* GI or GU cancers
* Severe Constipation in children only

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The investigators are collecting patients throughout North America (including the United States and Canada)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2006-01-15 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
observational study | through study completion, average of 10 years
  Outcome is candidate or causative genes for causing IC/BPS.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Brownstein, Ph.D., Principal Investigator — Boston Children's Hosptial
Locations (1):
- Boston Children's Hospital (BCH), Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from individual participants may be shared with other researchers. Other researchers will be approved by the internal review board at BCH.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: We will store data and samples indefinitely and may share samples/data with future collaborators.
Access Criteria: Data may be shared throughout the duration of the study. Collaborators will share de-identified data provided by study staff.

REFERENCES:
- [Background] Dimitrakov JD. A case of familial clustering of interstitial cystitis and chronic pelvic pain syndrome. Urology. 2001 Aug;58(2):281. doi: 10.1016/s0090-4295(01)01138-4. PMID 11489726
- [Result] Estrella E, Rockowitz S, Thorne M, Smith P, Petit J, Zehnder V, Yu RN, Bauer S, Berde C, Agrawal PB, Beggs AH, Gharavi AG, Kunkel L, Brownstein CA. Mendelian Disorders in an Interstitial Cystitis/Bladder Pain Syndrome Cohort. Adv Genet (Hoboken). 2022 Nov 27;4(1):2200013. doi: 10.1002/ggn2.202200013. eCollection 2023 Mar. PMID 36910591